CLINICAL TRIAL: NCT06771258
Title: What Effect Does Looking At Red Light Have on the Eye in Children and Young People? - a Proof-of-concept Study
Brief Title: Red Light Childhood Myopia Proof-of-concept
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: EDGE 166432
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intensity 1 (Active Comparator): Children will use red-light of the lowest intensity, twice daily for 3 minutes, at home
  Interventions: Other: Red Light (PDT)
- Intensity 2 (Active Comparator): Children will use red-light of low intensity, but slightly higher than in the Intensity 1 arm, twice daily for 3 minutes, at home
  Interventions: Other: Red Light (PDT)
- Intensity 3 (Active Comparator): Children will use red-light of medium intensity, slightly higher than in the Intensity 2 arm, twice daily for 3 minutes, at home
  Interventions: Other: Red Light (PDT)
- Intensity 4 (Active Comparator): Children will use red-light of medium intensity, slightly higher than in the Intensity 3 arm, twice daily for 3 minutes, at home
  Interventions: Other: Red Light (PDT)

INTERVENTIONS:
Other: Red Light (PDT) — Red LED light

SUMMARY:
In this project the research team will begin to find out whether shining a red LED light at the eyes can slow down the worsening of short-sightedness in children.

This is important, because short-sightedness now starts at a younger age and worsens faster than in the past. Many people are at risk of permanently losing their eyesight in middle-age because of short-sightedness.

The researchers plan to use red LED light, which is safe to use. Red-light treatment improves the blood flow at the back of the eye, in a layer called "choroid", which can be measured on eye-scans. The team have done a study with healthy adults, which showed that red-light is safe and gently improves the blood flow at the back of the eye. In adults, this has no effect on myopia, because their eyes are fully grown. In children, red-light may slow down myopia, and in this project, the researchers want to find out which level of red-light is needed to have this effect. The researchers will ask 24 children age 5-12 years to use red-light for three minutes twice a day for three months. Three will be 4 groups of children, and each group will use a different level of brightness. The researchers will measure the eye length and the thickness of the choroid at the start and 1 and 3 months later and compare the change in eye length between the different groups.

In practice, children will need to use the treatment for several years. The researchers will use the results of this study to prepare a longer study with more children.

ELIGIBILITY:
Inclusion Criteria:

* short-sightedness between -1.00D and -6.00 diopters in both eyes
* best-corrected visual acuity 0.1 logMAR or better in both eyes

Exclusion Criteria:

* underlying condition/syndrome causing myopia
* previous or current myopia-modifying treatment
* abnormal ocular refractive anatomy or previous intraocular or ocular surgery

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Axial length | 3 months
  The researchers will measure the length of the eyeballs using an optical biometer; these are the most sensitive outcome measure in myopia studies, and the least invasive measurement method.

SECONDARY OUTCOMES:
Spherical equivalent | 3 months
  The team will measure the refractive error (prescription for spectacles) using an open-view autorefractor, as a secondary measure of myopia progression.
Subfoveal choroidal thickness | 3 months
  The team will acquire an optical coherence tomography scan. On the scan, the researchers will measure the choroidal thickness, which is frequently used as a proxy measure of the treatment effect of interventions to slow myopia progression. The choroid is a vascular layer underneath the retina at the back of the eye.
Colour contrast sensitivity | 3 months
  As a safety measure, the researchers will measure colour contrast sensitivity on a computer-screen, showing participants coloured symbols on a grey background. This is the most sensitive test for photoreceptor health, the layer of cells in the retina which change light signals to electrical signals.
Visual acuity | 3 months
  As a secondary safety outcome, the researchers will measure the participant's visual acuity, using a test where participants read letters of reducing size on a chart.
Tolerability/usability | 3 months
  The researchers will ask participants open-ended questions about their thoughts and experience with using red-light treatment, and about easier ways for children to use it.

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Dahlmann-Noor, PhD, Principal Investigator — UCL
Locations (1):
- University College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided